CLINICAL TRIAL: NCT03502096
Title: The Influence of the Provision of a To-go Container on the Portion Size Effect in Women
Brief Title: Portion Size and To-go Container on Dinner Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jenny Craig, Inc. (Industry)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PortionSize105; R01DK059853 (NIH); NIFA Grant 2011-67001-30117 (Other Grant/Funding Number: United States Department of Agriculture)
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Eating Behavior
Keywords: portion size; food intake; energy intake; food choice
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The two factors were meal portion size and provision of a to-go container. The portion size factor was within-subjects (crossover). All subjects received each of the 4 portions served (the order in which portions were served was counterbalanced). The container factor was between-subjects. Subjects were randomly assigned to 1 of 2 groups: one group had uneaten food packaged to take home, the other group (control) did not.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100% portion size (Experimental): 100% portion sizes of all foods served (baseline). To-go container and controls received this meal.
  Interventions: Behavioral: To-Go container; Other: Control
- 125% portion size (Experimental): 125% of baseline portions served. To-go container and controls received this meal.
  Interventions: Behavioral: To-Go container; Other: Control
- 150% portion size (Experimental): 150% of baseline portions served. To-go container and controls received this meal.
  Interventions: Behavioral: To-Go container; Other: Control
- 175% portion size (Experimental): 175% of baseline portions served. To-go container and controls received this meal.
  Interventions: Behavioral: To-Go container; Other: Control

INTERVENTIONS:
Behavioral: To-Go container — Subjects were provided a to-go container in which leftover foods would be packaged
Other: Control — Subjects were not provided a to-go container with the meal

SUMMARY:
This study investigated whether the provision of a to-go container influenced the portion size effect at a meal. Following a screening visit, women came to the lab once a week for 4 weeks to eat a meal of multiple foods. At each visit, the portion size of the meal was varied in a counterbalanced order. Prior to their first meal, women were randomly assigned to one of two groups: a group that would have their leftovers packaged to go (to-go group) and a group that did not have leftovers packaged (control group). Women were instructed to eat ad libitum at the meals. They also answered questions about hunger and fullness as well as food characteristics before and after each meal. Following the final meal, subjects completed a series of questionnaires assessing subject characteristics as well as food characteristics. It was hypothesized that the effect of portion size on intake would be attenuated in subjects who received a to-go container with the meal. In addition, we aimed to identify any subject characteristics that moderated or exacerbated the portion size effect. It was also of interest to determine whether the portion size effect on individual foods were influenced by food characteristics such as perceived value.

ELIGIBILITY:
Inclusion Criteria:

* Regularly eats 3 meals/day
* Willing to avoid alcohol the day before and during test days
* Likes foods offered at test meals
* Body mass index 18 - 36 (kg/m*m)

Exclusion Criteria:

* Smokes
* Athlete in training
* Pregnant or breastfeeding
* Taking medication that may affect appetite or food intake
* Food allergies or dietary restrictions
* Currently have or recently been diagnosed with disease or disorder known to affect appetite

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 58 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in the weight of food consumed | Weeks 1, 2, 3, and 4
  Change in the weight of food consumed (in grams) across experimental conditions and intervention groups.
Change in energy intake | Weeks 1, 2, 3, and 4
  Change in energy intake (in kcal) across experimental conditions and intervention groups.

SECONDARY OUTCOMES:
Change in energy density consumed | Weeks 1, 2, 3, and 4
  Change in food energy density consumed (in kcal/g) across experimental conditions and intervention groups.
Change in intake of individual foods | Weeks 1, 2, 3, and 4
  Change in both the weight (g) and energy (kcal) consumed of individual foods served at the meal across experimental conditions and intervention groups.
Changes in post-meal measures of satiety | Weeks 1, 2, 3, and 4
  Changes in post-meal measures of satiety across experimental conditions and intervention groups using 100-mm visual analog scales.
Changes in post-meal ratings of meal characteristics | Weeks 1, 2, 3, and 4
  Changes in post-meal ratings of meal characteristics across experimental conditions and between subject groups using 100-mm visual analog scales.
Changes in ratings of food properties | Weeks 1, 2, 3, and 4
  Changes in post-meal ratings of food properties across experimental conditions and subject groups using 100-mm visual analog scales.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Rolls, PhD, Principal Investigator — The Pennsylvania State University